CLINICAL TRIAL: NCT00001888
Title: Asthma Sample Collection Protocol
Brief Title: Sample Collections From the Airways of Asthmatic Patients
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990076; 99-H-0076
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-22

CONDITIONS: Asthma
Keywords: Induced Sputum; Exhaled Breath Condensate; Fiberoptic Bronchoscopy; Bronchoscopy; mRNA; Natural History
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Asthmatics
- 2: Research Volunteers

SUMMARY:
Fiberoptic bronchoscopy is a procedure which involves passing a pencil-thin tube into the lung in order to collect fluid and cells from the airways. Fiberoptic bronchoscopy can collect cells from the walls of airways by gently brushing them (bronchial brushing). In addition, squirting small amounts of sterile water in to the airway and gently suctioning it back into the bronchoscope (bronchoalveolar lavage) collects cells.

In this study, researchers plan to perform these tests on patients with asthma and normal volunteers. This research may help to improve the understanding of the processes involved in airway inflammation and asthma.

DETAILED DESCRIPTION:
This tissue procurement protocol proposes to perform bronchoscopy with bronchoalveolar lavage, bronchial brushings, and bronchial wall biopsies, as well as to collect samples of sputum, exhaled breath condensates and blood, in order to evaluate the molecular mechanisms underlying the pathogenesis of airway inflammation, airway hyperresponsiveness, and airway remodeling in asthmatic subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

ASTHMATICS:

1. Patients undergoing a research bronchoscopy will be between 18 and 75 years of age, male or female. The diagnosis of asthma requires a history of intermittent, reversible expiratory flow limitation. In addition, patients will have demonstrated evidence of either an abnormal methacholine challenge or reversible airway obstruction. An abnormal methacholine challenge will be defined as a decrease in FEV1 of at least 20% at a PD20 dose < 200 microgram. Reversible airway obstruction will be defined as an improvement of at least 10% in either the FEV1 or FVC following bronchodilator treatment. Methacholine challenge testing will not be performed if the subject has a history of allergy to methacholine. Results of testing performed by the subject s primary care provider may be accepted as evidence of reversible airflow obstruction.
2. For women of childbearing potential, negative pregnancy test and willingness to adhere to reliable birth control methods prior to

   bronchoscopy or sputum induction.
3. Asthmatic research subjects who will only be providing research blood specimens, nasal epithelial lining fluid, spontaneously expectorated sputum, or exhaled breath condensate, and will not be undergoing a research bronchoscopy or sputum induction, may participate in the protocol by providing a clinical history that they have asthma and are not pregnant. Documentation of an abnormal methacholine challenge or reversible airflow obstruction or a negative pregnancy test, for women of childbearing age, will not be required for donation of research blood specimens, or other non-invasive samples, such as nasal epithelial lining fluid, sputum, or exhaled breath condensate.

EXCLUSION CRITERIA:

ASTHMATICS:

Diagnosis of a pulmonary disorder other than asthma (e.g., chronic bronchitis, cystic fibrosis, HIV-related lymphocytic airway inflammation).

History of drug or alcohol abuse within the past year.

Positive test for human immunodeficiency virus (to exclude patients with HIV-related lymphocytic airway inflammation) or hepatitis virus.

INCLUSION CRITERIA - RESEARCH VOLUNTEERS:

1. Research volunteers undergoing a research bronchoscopy will be between 18 and 75 years of age, male or female.
2. A negative inhalational methacholine challenge as defined by the absence of a 20% decrease in FEV1 at a PD20 dose of > 400 microgram (normal bronchial hyperresponsiveness). Methacholine challenge testing will not be performed if the subject has a history of allergy to methacholine. Results of testing performed by the subject s primary care provider may be accepted as evidence of a negative methacholine challenge.
3. For women of childbearing potential, negative pregnancy test within 2 weeks prior to bronchoscopy and willingness to adhere to reliable birth control methods prior to bronchoscopy or sputum induction.
4. Research volunteers who will only be providing research blood specimens, nasal epithelial lining fluid, sputum, spontaneously expectorated sputum, or exhaled breath condensate, and will not be undergoing a research bronchoscopy or sputum induction, may be included in the protocol without documentation of a negative inhalational methacholine challenge or a negative pregnancy test if they provide a history that they do not have asthma and that they are not currently pregnant, for women of childbearing age.

EXCLUSION CRITERIA - RESEARCH VOLUNTEERS:

Same as the asthmatic exclusion criteria plus a history of asthma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual between the ages of 18 and 75 with asthma will be accepted into the study. Since asthma has a roughly equivalent prevalence in groups differing in race and gender, recruitment of study participants will be aimed at selecting a study population which reflect this diversity. Asthmatic or research volunteers with HIV infection will be excluded from the study so as not to include patients with HIV-related lymphocytic airway inflammation. Volunteers will be obtained through the NIH Clinical Research Volunteer Program or other standard channels at NIH.
Sampling Method: Non-Probability Sample
Enrollment: 574 (Actual)
Dates: Start 1999-06-02 (Actual)

PRIMARY OUTCOMES:
Assess the role of apolipoprotein and lipid pathways in asthmatic and non-asthmatic subjects. | ongoing
  These studies will increase the understanding of the pathogenic mechanisms underlying asthmatic airway inflammation and may identify novel therapeutic targets.

SECONDARY OUTCOMES:
Assess the role of exosome-associated proteins and receptors in the regulation of airway inflammatory responses | ongoing
  These studies will increase the understanding of the pathogenic mechanisms underlying asthmatic airway inflammation and may identify novel therapeutic targets.
Assess the expression, regulation, and function of differentially expressed proteins and genes in human airway structural and inflammatory cell populations in asthma | ongoing
  These studies will increase the understanding of the pathogenic mechanisms underlying asthmatic airway inflammation and may identify novel therapeutic targets.
Assess the relative contribution of specific soluble pro-inflammatory cytokines and receptors in asthmatic bronchoalveolar lavage fluid (BALF) in mediating airway structural and inflammatory cell responses | ongoing
  These studies will increase the understanding of the pathogenic mechanisms underlying asthmatic airway inflammation and may identify novel therapeutic targets.
Assess the expression, regulation, and function of proteins regulating the release of soluble receptors and mediators from asthmatic inflammatory and structural cell populations | ongoing
  These studies will increase the understanding of the pathogenic mechanisms underlying asthmatic airway inflammation and may identify novel therapeutic targets.

CONTACTS AND LOCATIONS:
Overall Officials: Amisha V Barochia, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yao X, Kaler M, Qu X, Kalidhindi RSR, Sviridov D, Dasseux A, Barr E, Keeran K, Jeffries KR, Yu ZX, Gao M, Gordon S, Barochia AV, Mills J, Shahid S, Weir NA, Kalchiem-Dekel O, Theard P, Playford MP, Stylianou M, Fitzgerald W, Remaley AT, Levine SJ. Asthmatic patients with high serum amyloid A have proinflammatory HDL: Implications for augmented systemic and airway inflammation. J Allergy Clin Immunol. 2024 Apr;153(4):1010-1024.e14. doi: 10.1016/j.jaci.2023.11.917. Epub 2023 Dec 12. PMID 38092139
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-H-0076.html